CLINICAL TRIAL: NCT04193553
Title: A Multicentre, Comparative, Placebo-controlled, Double-blinded, Phase II Study of the Efficacy of Lenvatinib in Patients With Locally Advanced or Metastatic GIST After Failure of Imatinib and Sunitinib
Brief Title: Multicentre Placebo-controlled Double-blinded Phase II Study of Lenvatinib Efficacy in Patients With Locally Advanced or Metastatic GIST (Gastrointestinal Stromal Tumor) After Imatinib/Sunitinib Failure
Acronym: LENVAGIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ET18-291 - LENVAGIST
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-04

CONDITIONS: Gastro Intestinal Stromal Tumour
Keywords: Gastro Intestinal Stromal Tumour; Locally advanced or metastatic; Tyrosine kinase inhibitors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenvatinib + Best Supportive Care (Experimental)
  Interventions: Drug: Lenvatinib; Other: Best supportive care
- Placebo + Best Supportive Care (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Best supportive care

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administered continuously but patient's follow-up visits will be scheduled monthly.
  The starting dose of study treatment is 24mg, once daily, at the same time. Recommendations for dose reductions will be respected according to BI Lenvatinib.
  If a patient misses a dose, and it cannot be taken within 12 hours, then that dose should be skipped and the next dose should be taken at the usual time of administration.
  Study treatments will be continued until a treatment discontinuation criteria is met.
  Arms: Lenvatinib + Best Supportive Care
Drug: Placebo — Placebo will be administered continuously but patient's follow-up visits will be scheduled monthly.
  The starting dose of study treatment is 24mg, once daily, at the same time. Recommendations for placebo dose reductions are the same as for Lenvatinib. If a patient misses a dose, and it cannot be taken within 12 hours, then that dose should be skipped and the next dose should be taken at the usual time of administration.
  Study treatments will be continued until a treatment discontinuation criteria is met.
  In case disease progression, patients in control arm could switch in the Lenvatinib + BSC arm.
  Arms: Placebo + Best Supportive Care
Other: Best supportive care — At any time during the study, patients should receive best supportive care. Best Supportive care as medically indicated for the patient's well-being may be prescribed at the investigator's discretion. Based on the patient's condition, it may consist (but not limited) of analgesics, antibiotics, steroids, blood transfusion, antiemetics, antidepressants/anxiolytics, nutritional counselling, psychological support, palliative radiotherapy…

SUMMARY:
The primary objective is to compare the efficacy of lenvatinib plus Best Supportive Care versus Placebo plus Best Supportive Care in the treatment of patients with advanced GIST, after failure of imatinib and sunitinib.

DETAILED DESCRIPTION:
Even though the prognosis of advanced GIST has been tremendously improved by the introduction of tyrosine kinase inhibitors, the vast majority of patients will develop secondary resistance to these agents.

The therapeutic options of patients with advanced GIST with resistance (or intolerance) to imatinib and sunitinib remain then very limited and prognosis of patients are very poor.

Nilotinib has an inferior activity in first line setting as compared to imatinib. Sorafenib has been evaluated in off-label and compassionate use studies with a median PFS close to 3 to 4 months, and a median overall survival close to 9 months with few prolonged tumor control and limited availability.

Regorafenib was tested in a phase II and a randomized phase III trial (GRID) in this setting , and provided a significant PFS advantage with no significant improvement in OS.

There are no recognized standard options in patients whose tumors progress after 3 or more TKIs. The recently updated guidelines from ESMO in 2014, included the reintroduction of imatinib in an attempt to control the progression of the sensitive cell clones, and on the basis of the results of the RIGHT study.

This is therefore a situation with a clear unmet medical need.

Lenvatinib is a broad spectrum TKI targeting oncogenes KIT and RET and receptor tyrosine kinases, PDGFRA, VEGFR 1-3 and FGFR 1-4. It has demonstrated activity in iodine resistant metastatic thyroid cancers. Whether lenvatinib would be a useful agent in patients with GIST is not known but there is a rationale to investigate its activity in patients with advanced GIST.

In the present study, we propose to analyze the antitumor activity of lenvatinib in patients with GIST failing to at least imatinib and sunitinib in a randomized setting, vs placebo.

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female ≥ 18 years at the day of consenting to the study.

I2. Patient must have histologically confirmed diagnosis of GIST.

I3. Disease must be locally advanced or metastatic.

I4. Patient who failed (disease progression and/or intolerance) previously at least to imatinib and sunitinib.

Nota Bene: patients with more than 2 previous anticancer treatments are eligible.

I5. Patient must have evidence of measurable disease as per the RECIST version 1.1 (Appendix 2).

I6. Patient must have documented disease progression. I7. ECOG performance status 0, 1 or 2 (Appendix 3).

I8. Patient must have normal organ and bone marrow function as defined below:

* Hematologic

  * Absolute neutrophil count (ANC) ≥ 1.5 Gi/L
  * Haemoglobin ≥ 9 g/dl (5.6 mmol/l) (subjects may not have had a transfusion within 7 days of screening assessment)
  * Platelets ≥ 100 Gi/l
* Coagulation panel

  * Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.2 X upper limit of normal (ULN)
  * Partial thromboplastin time (PTT) ≤ 1.2 X ULN Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
* Hepatic

  * Total bilirubin ≤ 1.5 X ULN
  * AST and ALT ≤ 2.5 X ULN
* Renal

  * Serum creatinine ≤ 1.5 mg/dl (133 µmol/l) Or, if greater than 1.5 mg/dl: calculated creatinine clearance ≥ 50 ml/min
  * Urine Protein to Creatinine ratio (UPC) < 1; If UPC > 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1g.

I9. Patient and his/her partner using an effective contraception as defined in Appendix 1.

I10. Patient able to understand and willingness for follow-up visits. I11. Patient covered by a medical insurance. I12. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to any study-specific procedure.

Exclusion Criteria:

E1. Patient with a documented mutation in PDGFRA exon 18 (D842V substitution).

E2. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

* Active peptic ulcer disease
* Known intraluminal metastatic lesions with risk of bleeding
* Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:
* Malabsorption syndrome
* Major resection of the stomach or small bowel.

E3. Any active/uncontrolled infection, including known infection with HIV, Hepatitis B or Hepatitis C.

E4. Corrected QT interval (QTc) > 480 msecs using Bazett's formula

E5. History of any one or more of the following cardiovascular conditions within the past 6 months prior to the first dose of study drug:

* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery bypass graft surgery
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) classification.

E6. Poorly controlled arterial hypertension (Systolic blood pressure: 150mmHg / Diastolic blood pressure: 90mmHg).

Note: Patients with high blood pressure can be enrolled provided that the hypertension is well controlled at a stable dose of antihypertensive therapy for at least 1 week prior to lenvatinib start).

E7. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).

E8. Evidence of active bleeding or bleeding diathesis. E9. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.

E10. Clinically significant haemoptysis within 8 weeks of first dose of study drug.

E11. Any serious and/or unstable pre-existing medical, psychiatric, or other condition (geographic, social…) that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

E12. Unable or unwilling to discontinue use of prohibited medications list in Section 6.3 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.

E13. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.

E14. Inability to swallow E15. Any contraindication to Lenvima®, according to its Summary of Product Characteristics E16. History of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition of lenvatinib E17. Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results.

E18. Pregnant or breastfeeding women. Women of childbearing potential (Appendix 1) are required to have a negative serum pregnancy test within 72 hours prior to study treatment start. A positive urine test must be confirmed by a serum pregnancy test Note: Female if applicable, subjects should discontinue breast-feeding prior to the first dose of study drug and should refrain from breastfeeding throughout the treatment period and for 14 days following the last dose of study drug.

E19. Patient under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 30 months
  PFS, defined as the time from the date of randomisation to the date of the first documented radiological progression (RECIST 1.1) or death due to any cause.
  PFS will be estimated using the Kaplan-Meier method and will be described in terms of median PFS per arm, and hazard ratio for progression between the 2 arms. Associated 2-sided 95% CI for the estimates will be provided.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 30 months
  OS, is defined as the time from the date of randomisation until the date of death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Objective Response Rate (ORR) for patient in the blinded part of the study | Up to 30 months
  ORR, is the proportion of patients with a Complete Response or Partial Response as Best Overall Response.
Best Overall Response (BOR) for patient in the blinded part of the study | Up to 30 months
  BOR, is described as the proportion of patients with a best overall response of Complete Response, Partial Response, Stable Disease or Progressive Disease.
Quality of Life (QoL) for patient in the blinded part of the study | Up to 30 months
  QoL, will be assessed using the EORTC QLQ-C30. Scores will be calculated at each time point according to the scoring manuals. Descriptive statistics will be used to evaluate baseline scores and evolution of scores from baseline to each time point. Data will be compared between arms using the Student's t-test.
Patient's tolerance to treatment | Up to 30 months
  The safety will be described mainly on the frequency of adverse events coded using the common toxicity criteria (NCI-CTCAE v5.0) grade. Descriptive statistics will be provided for characterizing and assessing patient tolerance to treatment. Adverse events will be coded according to the MedDRA®.
Progression-Free Survival (PFS) In patients from the placebo arm who switched into the active treatment group | Up to 30 months
  OS, is defined as the time from the date of randomisation until the date of death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.

OTHER OUTCOMES:
Mutation profile : KIT | Inclusion
  Determined by immunohistochemistry (archival formalin fixed paraffin embedded tumor sample)
Mutation profile: PDGFR | Inclusion
  Determined by immunohistochemistry (archival formalin fixed paraffin embedded tumor sample)
Pharmacokinetic properties of lenvatinib for patient in the blinded part of the study | Inclusion, Day 1 of cycles 2, 3, 4, 5, up to 12 months (28 days cycle)
  Trough levels of lenvatinib

CONTACTS AND LOCATIONS:
Overall Officials: Axel LE CESNE, Ph, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (14):
- France (14):
  - Centre Antoine LACASSAGNE, Nice, Alpes-Maritimes
  - Hopital de La Timone, Marseille, Bouches Du Rhône
  - Institut Paoli Calmette, Marseille, Bouches-du-Rhône
  - Centre Georges-François Leclerc, Dijon, Bourgogne-Franche-Comté
  - Institut Bergonié, Bordeaux, Gironde
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse, Haute-Garonne
  - Centre Oscar LAMBRET, Lille, Hauts-de-France
  - Centre Eugène Marquis, Rennes, Ille-et-Vilaine
  - ICO Centre René Gauducheau, Saint-Herblain, Loire-Atlantique
  - CHU de Reims, Reims, Marne
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Léon Bérard, Lyon, Rhône
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - CHU Poitiers, Poitiers, Vienne